CLINICAL TRIAL: NCT02921061
Title: Phase 1/2 Study of Concurrent Decitabine in Combination With G-CSF, Cladribine, Cytarabine, and Mitoxantrone (G-CLAM) in Adults With Newly Diagnosed Acute Myeloid Leukemia (AML) or High-Risk Myelodysplastic Syndromes (MDS)
Brief Title: Decitabine With GCLAM for Adults With Newly Diagnosed, Relapsed, or Refractory AML or High-Risk MDS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9713; NCI-2016-01401 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9713 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH); RG9216023 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2016-09-29; First posted 2016-09-30 (Estimated); Results first posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-01

CONDITIONS: Mixed Phenotype Acute Leukemia; Previously Treated Myelodysplastic Syndrome; Recurrent Adult Acute Myeloid Leukemia; Recurrent High Risk Myelodysplastic Syndrome; Refractory Acute Myeloid Leukemia; Refractory High Risk Myelodysplastic Syndrome; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Biphenotypic, Acute; Leukemia, Myeloid, Acute | interventions — Cladribine; Cytarabine; Decitabine; Injections; Filgrastim; Granulocyte Colony-Stimulating Factor; Mitoxantrone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | US Export: Yes

ARMS (1):
- Treatment (decitabine, G-CLAM) (Experimental): INDUCTION: Patients receive decitabine IV over 1 hour on days 1-10. Patients also receive filgrastim SC on days 0-5, cladribine IV over 2 hours on days 1-5, cytarabine IV over 2-4 hours on days 1-5, and mitoxantrone hydrochloride IV over 60 minutes on days 1-3.
  RE-INDUCTION: Patients who do not achieve MRDneg CR after first induction are eligible for re-induction. Patients receive the same treatment as during induction except that decitabine is omitted.
  CONSOLIDATION THERAPY: Beginning 6 weeks after achieving MRDneg CR or CR/CR with CRi after induction and/or re-induction, patients are eligible to receive filgrastim, cladribine, and cytarabine as in Induction. Treatment may be repeated for up to 4 courses in the absence of disease progression or unacceptable toxicity. Subsequent consolidation cycles would be given after recovery from the previous cycle (roughly 4-6 weeks).
  Interventions: Drug: Cladribine; Drug: Cytarabine; Drug: Decitabine; Biological: Filgrastim; Other: Laboratory Biomarker Analysis; Drug: Mitoxantrone Hydrochloride

INTERVENTIONS:
Drug: Cladribine — Given IV
  Other Names: 2-CdA; 2CDA; CdA; Cladribina; Leustat; Leustatin; Leustatine; RWJ-26251
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Decitabine — Given IV
  Other Names: 5-Aza-2'-deoxycytidine; Aza-TdC; Dacogen; Decitabine for Injection; Deoxyazacytidine; Dezocitidine
Biological: Filgrastim — Given SC
  Other Names: FILGRASTIM, LICENSE HOLDER UNSPECIFIED; G-CSF; Neupogen; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; rG-CSF; Tevagrastim
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Mitoxantrone Hydrochloride — Given IV
  Other Names: CL 232315; DHAD; DHAQ; Dihydroxyanthracenedione Dihydrochloride; Mitoxantrone Dihydrochloride; Mitoxantroni Hydrochloridum; Mitozantrone Hydrochloride; Mitroxone; Neotalem; Novantrone; Onkotrone; Pralifan

SUMMARY:
This phase I/II trial studies the side effects and best dose of decitabine when given together with filgrastim, cladribine, cytarabine, and mitoxantrone hydrochloride in treating patients with acute myeloid leukemia or myelodysplastic syndrome that is newly diagnosed, has come back or has not responded to treatment. Drugs used in chemotherapy, such as decitabine, cladribine, cytarabine, and mitoxantrone hydrochloride work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Colony-stimulating factors, such as filgrastim, may increase the production of blood cells and may help the immune system recover from the side effects of chemotherapy. Decitabine, filgrastim, cladribine, cytarabine, and mitoxantrone hydrochloride may work better in treating patients with acute myeloid leukemia and myelodysplastic syndrome.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Estimate the maximum tolerated dose (MTD) of decitabine when used concomitantly with filgrastim, cladribine, cytarabine, and mitoxantrone hydrochloride (G-CLAM) in patients with newly diagnosed acute myeloid leukemia (AML) and high-risk myelodysplastic syndrome (MDS).

II. Compare, within the limits of a phase 1/2 study, the rate of complete remission without measurable residual disease (minimal residual disease negative [MRDneg] complete remission [CR]) with decitabine + G-CLAM at the MTD compared to similar patients treated previously with G-CLAM alone.

SECONDARY OBJECTIVES:

I. Evaluate, within the limits of a phase 1/2 study, disease response (complete remission, overall response rate) relapse-free survival (RFS), event-free survival (EFS), and overall survival (OS) in patients with newly-diagnosed AML / high-risk MDS.

II. Describe, within the limits of a phase 1/2 study, the toxicity profile of the study regimen.

OUTLINE: This is a dose de-escalation study of decitabine.

INDUCTION: Patients receive decitabine intravenously (IV) over 1 hour on days 1-10. Patients also receive filgrastim subcutaneously (SC) on days 0-5, cladribine IV over 2 hours on days 1-5, cytarabine IV over 2-4 hours on days 1-5, and mitoxantrone hydrochloride IV over 60 minutes on days 1-3.

RE-INDUCTION: Patients who do not achieve MRDneg CR after first induction are eligible for re-induction. Patients receive the same treatment as during induction except that decitabine is omitted.

CONSOLIDATION THERAPY: Beginning 6 weeks after achieving MRDneg CR or CR/CR with incomplete count recovery (CRi) after induction and/or re-induction, patients are eligible to receive filgrastim, cladribine, and cytarabine as in Induction. Treatment may be repeated for up to 4 courses in the absence of disease progression or unacceptable toxicity. Subsequent consolidation cycles would be given after recovery from the previous cycle (roughly 4-6 weeks).

After completion of study treatment, patients are followed up at for 1 month and every 3 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* For patients with newly diagnosed disease: diagnosis of "high-grade" MDS (>= 10% blasts by morphology) or AML other than acute promyelocytic leukemia (APL) with t(15;17)(q22;q12) or variants according to the 2016 World Health Organization (WHO) classification; for patients with relapsed/refractory disease: prior diagnosis of "high-risk" MDS or non-APL AML, with relapsed/refractory disease according to 2003 recommendations of the International Working Group, requiring first or subsequent salvage therapy; patients with mixed phenotype acute leukemia (MPAL) are eligible
* Outside diagnostic material is acceptable as long as peripheral blood and/or bone marrow slides are reviewed at the study institution; flow cytometric analysis of peripheral blood and/or bone marrow should be performed according to institutional practice guidelines
* Patients with prior autologous or allogeneic hematopoietic cell transplantation (HCT) are eligible if relapse occurs provided symptoms of graft-versus host disease are well controlled with stable use of immunosuppressive agents
* Treatment-related mortality (TRM) score =< 9.2 as calculated with simplified model
* Should be off any active therapy for AML with the exception of hydroxyurea for at least 14 days prior to study registration unless patient has rapidly progressive disease, and all grade 2-4 non-hematologic toxicities should have resolved
* May have previously received monotherapy with demethylating agents for MDS or AML or treatment with a mitoxantrone- or cladribine-based regimen for MDS or AML, including G-CLAM, but not demethylating agent as priming for or in combination with chemotherapy
* Patients with symptoms/signs of hyperleukocytosis or white blood cells (WBC) > 100,000/uL can be treated with leukapheresis or may receive up to 2 doses of cytarabine (up to 500 mg/m^2/dose) prior to enrollment
* Bilirubin =< 2.5 x institutional upper limit of normal (IULN) unless elevation is thought to be due to hepatic infiltration by AML, Gilbert's syndrome, or hemolysis (assessed within 14 days prior to registration)
* Serum creatinine =< 2.0 mg/dL (assessed within 14 days prior to registration)
* Left ventricular ejection fraction >= 45%, assessed within 3 months prior to registration, e.g. by multigated acquisition scan (MUGA) scan or echocardiography, or other appropriate diagnostic modality and no clinical evidence of congestive heart failure; if the patient had anthracycline-based therapy since the most recent cardiac assessment, cardiac evaluation should be repeated if there is clinical or radiographic suspicion of cardiac dysfunction, or if the previous cardiac assessment was abnormal
* Women of childbearing potential and men must agree to use adequate contraception
* Ability to understand and willingness to sign a written consent

Exclusion Criteria:

* Myeloid blast crisis of chronic myeloid leukemia (CML), unless patient is not considered candidate for tyrosine kinase inhibitor treatment
* Concomitant illness associated with a likely survival of < 1 year
* Active systemic fungal, bacterial, viral, or other infection, unless disease is under treatment with anti-microbials and/or controlled or stable (e.g. if specific, effective therapy is not available/feasible or desired [e.g. chronic viral hepatitis, human immunodeficiency virus (HIV)]); patient needs to be clinically stable as defined as being afebrile and hemodynamically stable for 24-48 hours
* Known hypersensitivity to any study drug
* Pregnancy or lactation
* Patients may not be receiving any other investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-11-17 (Actual); Primary Completion 2018-10-24 (Actual); Study Completion 2018-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roland Walter, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

REFERENCES:
- [Derived] Palmieri R, Buckley SA, Othus M, Halpern AB, Percival MM, Scott BL, Hendrie PC, Becker PS, Oehler VG, Estey EH, Walter RB. Randomized phase 1 study of sequential ("primed") vs. concurrent decitabine in combination with cladribine, cytarabine, G-CSF, and mitoxantrone (CLAG-M) in adults with newly diagnosed or relapsed/refractory acute myeloid leukemia (AML) or other high-grade myeloid neoplasm. Leuk Lymphoma. 2020 Jul;61(7):1728-1731. doi: 10.1080/10428194.2020.1728754. Epub 2020 Feb 20. No abstract available. PMID 32077361

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Though this is a dose escalation study, all patients ultimately received decitabine at the same dose (20 mg/m2) and the same additional drugs (G-CLAM) over the same dosing schedule.
Groups:
- Treatment (Decitabine 20 mg/m2 and G-CLAM): Patients receive induction therapy comprising decitabine IV over 1 hour (20 mg/m2) on days 1-10 and G-CLAM (filgrastim SC on days 0-5, cladribine IV over 2 hours on days 1-5, cytarabine IV over 2-4 hours on days 1-5, and mitoxantrone IV over 60 minutes on days 1-3).
  Patients who do not achieve MRDneg CR after first induction are eligible for re-induction with G-CLAM.
  Beginning 6 weeks after achieving MRDneg CR or CR/CR with CRi after induction and/or re-induction, patients are eligible to receive consolidation therapy comprising GLCA (filgrastim, cladribine, cytarabine) for up to 4 cycles. Subsequent consolidation cycles would be given after recovery from the previous cycle (roughly 4-6 weeks).
Period: Overall Study
Arm/Group | Treatment (Decitabine 20 mg/m2 and G-CLAM)
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Decitabine 20 mg/m2 and G-CLAM)
Number analyzed (Participants) | 28
Age, Continuous [Median (Full Range); unit: years] | 67 [28 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 25
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Dose Limiting Toxicities (DLTs) at the Maximum Tolerated Dose (MTD) for Decitabine When Given Together With G-CLAM Toxicities (DLTs) (Phase I)
Description: Evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0. MTD is defined as the highest dose studied in which the incidence of DLT is < 33%. Each participant was monitored for DLTs in the first 20 days of treatment. DLTs monitored included
  1. any grade 3 non-hematologic toxicity lasting more than 48 hours that resulted in more than a 7 day delay of the subsequent treatment cycle (except for febrile neutropenia or infection)
  2. any grade 4 or greater non-hematologic toxicity (except febrile neutropenia and infection unless a direct consequence of a treatment-related toxicity, and except constitutional symptoms if they recovered to grade 2 or less within 14 days)
  3. lack of recovery of the absolute neutrophil count to 500/microliter or greater and lack of self-sustained platelet count of at least 50,000/microliter by treatment day +49 with no evidence of residual leukemia
Time Frame: Up to 49 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Decitabine 20 mg/m2 and G-CLAM)
Number analyzed (Participants) | 28
Participants | 3

2. Secondary Outcome: Number of Participants With Minimal Residual Disease Negative (MRDneg) Complete Remission (Phase II)
Description: Compared to historical controls of filgrastim, cladribine, cytarabine, and mitoxantrone hydrochloride (G-CLAM) alone. A Simon Minimax two-stage design will be used.
Time Frame: Up to 1 year
Measure: Number; unit: participants
Arm/Group | Treatment (Decitabine 20 mg/m2 and G-CLAM)
Number analyzed (Participants) | 28
participants | 13

3. Secondary Outcome: Number of Participants Who Achieved Remission (Complete Remission [CR]/CR With Incomplete Peripheral Blood Count Recovery [CRi])
Time Frame: Up to 1 year
Measure: Number; unit: participants
Arm/Group | Treatment (Decitabine 20 mg/m2 and G-CLAM)
Number analyzed (Participants) | 28
participants | 13

4. Secondary Outcome: Number of Participants With Overall Survival
Time Frame: Up to 1 year
Measure: Number; unit: participants
Arm/Group | Treatment (Decitabine 20 mg/m2 and G-CLAM)
Number analyzed (Participants) | 28
participants | 9

5. Secondary Outcome: Number of Participants With Relapse-free Survival
Time Frame: Up to 1 year
Measure: Number; unit: participants
Arm/Group | Treatment (Decitabine 20 mg/m2 and G-CLAM)
Number analyzed (Participants) | 28
participants | 8

6. Secondary Outcome: Number of Participants With Event-free Survival
Time Frame: Up to 1 year
Measure: Number; unit: participants
Arm/Group | Treatment (Decitabine 20 mg/m2 and G-CLAM)
Number analyzed (Participants) | 28
participants | 8

ADVERSE EVENTS:
Time Frame: All-Cause Mortality assessed for up to 12 months; Serious and Other Adverse Events assessed for up to 1 month after treatment duration of about 10 days concluded
Arm/Group | Treatment (Decitabine 20 mg/m2 and G-CLAM)
All-Cause Mortality (participants affected / at risk) | 19/28
Serious Adverse Events (participants affected / at risk) | 2/28
Other Adverse Events (participants affected / at risk) | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Decitabine 20 mg/m2 and G-CLAM) (N=28)
Sepsis (Infections and infestations) | 1
Cardiogenic shock/heart failure (Cardiac disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Decitabine 20 mg/m2 and G-CLAM) (N=28)
acute kidney injury, grade 3 (Renal and urinary disorders) | 1
aortic valve disease, grade 3 (Cardiac disorders) | 1
AST increased, grade 3 (Hepatobiliary disorders) | 1
atrial fibrillation, grade 3 (Cardiac disorders) | 2
atrial fibrillation, grade 4 (Cardiac disorders) | 1
back pain, grade 3 (General disorders) | 1
delirium, grade 3 (Psychiatric disorders) | 1
diarrhea, grade 3 (Gastrointestinal disorders) | 2
duodenal hemorrhage, grade 4 (Gastrointestinal disorders) | 1
dyspnea, grade 4 (Respiratory, thoracic and mediastinal disorders) | 1
encephalopathy, grade 4 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
fatigue, grade 3 (General disorders) | 1
febrile neutropenia, grade 3 (Infections and infestations) | 27
hyperbilirubinemia, grade 4 (Blood and lymphatic system disorders) | 1
hypertension, grade 3 (General disorders) | 2
hypokalemia, grade 3 (Metabolism and nutrition disorders) | 2
hypotension, grade 3 (General disorders) | 1
hypoxemia, grade 3 (General disorders) | 7
infective endocarditis, grade 3 (Cardiac disorders) | 1
LV systolic dysfunction, grade 4 (General disorders) | 1
maculopapular rash, grade 3 (Skin and subcutaneous tissue disorders) | 1
myocardial infarction, grade 4 (Cardiac disorders) | 1
nausea, grade 3 (General disorders) | 1
phlebitis infective, grade 3 (Vascular disorders) | 1
pleural effusions, grade 3 (Respiratory, thoracic and mediastinal disorders) | 1
pulmonary nodules, grade 3 (Respiratory, thoracic and mediastinal disorders) | 7
sinusitis, grade 3 (General disorders) | 1
syncope, grade 3 (General disorders) | 3
tumor lysis syndrome, grade 3 (General disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-10): https://cdn.clinicaltrials.gov/large-docs/61/NCT02921061/Prot_SAP_000.pdf